CLINICAL TRIAL: NCT05963620
Title: Long-term Follow-up of a Randomized Comparison of Percutaneous Coronary Intervention Versus Coronary Artery Bypass Surgery in Unprotected Left Main Disease
Brief Title: Long-term Follow-up of a Randomized Comparison of Percutaneous Coronary Intervention Versus Coronary Artery Bypass Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0444
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Coronary Stenosis; Coronary Artery Disease
Keywords: Percutaneous coronary intervention; sirolimus-eluting stent; coronary artery bypass grafting
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- percutaneous coronary intervention (PCI): percutaneous coronary intervention (PCI) with sirolimus-eluting stents
  Interventions: Other: percutaneous coronary intervention vs bypass graft surgery
- coronary artery bypass grafting (CABG): coronary artery bypass graft surgery
  Interventions: Other: percutaneous coronary intervention vs bypass graft surgery

INTERVENTIONS:
Other: percutaneous coronary intervention vs bypass graft surgery — retrieve long term follow up data on clinical outcome of study population, no intervention

SUMMARY:
This is a long-term follow-up of a completed clinical trial which compared percutaneous coronary intervention (PCI) using sirolimus-eluting stents and coronary artery bypass grafting (CABG) in patients with unprotected left main coronary artery disease.

The purpose of the study is to obtain retrospective long-term data on clinical outcome of the study population.

DETAILED DESCRIPTION:
The randomized multicenter, open-label trial "Percutaneous Coronary Intervention (PCI) With Drug-Eluting Stents (DES) Versus Coronary Artery Bypass Graft (CABG) for Patients With Significant Left Main Stenosis" was conducted at 4 tertiary care centers in Germany. 201 patients with unprotected left main stem stenosis (≥50%) with or without additional multivessel coronary artery disease were enrolled in a 1:1 ratio from July 2003 through February 2009. Results were published: https://pubmed.ncbi.nlm.nih.gov/21272743/

Long-term follow-up will be performed by a structured telephone interview using a standardized questionnaire by an interviewer blinded to treatment allocation. Wherever possible, data will be completed and verified by health care records. Retrospective data of the underlying randomized study will be included in data analysis.

ELIGIBILITY:
Inclusion Criteria:

* alive participants of underlying study who give their consent to participate
* deceased participants of underlying study

Exclusion Criteria:

* alive participants of underlying study who do not consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants of the preceding study: Percutaneous Coronary Intervention (PCI) With Drug-Eluting Stents (DES) Versus Coronary Artery Bypass Graft (CABG) for Patients With Significant Left Main Stenosis
Sampling Method: Non-Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
All-cause death | approximately 15 years after procedure
  further categorized into cardiovascular, noncardiovascular, and undetermined deaths

SECONDARY OUTCOMES:
composite secondary endpoint | approximately 15 years after procedure
  all-cause death, myocardial infarction or repeat target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Desch, MD, Study Chair — Heart Center Leipzig at University of Leipzig
Locations (4):
- Germany (4):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen, Baden Würtemberg
  - Klinikum der Ludwig-Maximilians Universität München, München, Bavaria
  - München Klinik Neuperlach, München, Bavaria
  - Heart Center Leipzig at University of Leipzig, Leipzig, Saxony